CLINICAL TRIAL: NCT04318704
Title: An Open Label Study of the Efficacy, Safety and Tolerability of NP-120 on Idiopathic Pulmonary Fibrosis and Its Associated Cough
Brief Title: Efficacy, Safety and Tolerability of NP-120 on Idiopathic Pulmonary Fibrosis and Its Associated Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Algernon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGN120-1
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Cough
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough | interventions — ifenprodil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Active (Other): Ifenprodil
  Interventions: Drug: Ifenprodil

INTERVENTIONS:
Drug: Ifenprodil — Ifenprodil 20 mg TID

SUMMARY:
NP-120 (Ifenprodil) has been shown to mediate anti-inflammatory responses and reduce pulmonary fibrosis in a murine model of Idiopathic Pulmonary Fibrosis (IPF). In addition, NP-120 significantly reduced both cough frequency and onset in a guinea pig tussive model. The purpose of this proof-of-concept trial is to determine the efficacy of NP-120 in the treatment of IPF and its associated cough.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with a diagnosis of IPF established during the previous seven years according to ATS/ERS/Fleischner criteria.
2. Score ≥ 40 mm on the Cough Severity VAS at Screening
3. Lung function parameters as follows:

   1. Forced Vital Capacity (FVC) ≥ 45% of the predicted value at screening.
   2. Diffusion lung capacity for carbon monoxide (DLCO) (corrected for Hb) of 30% to 79% of the predicted value at screening.
4. Any existing Standard of Care (SoC) treatment (e.g. pirfenidone or nintedanib) must be deemed as stable (minimum three months) before enrollment.
5. Subjects must sign and date a written, informed consent form and any required authorization prior to initiation of any study procedures.

Exclusion Criteria:

1. Currently has significant airways obstruction: Forced Expiratory Volume in 1 s (FEV1)/Forced Vital Capacity (FVC) ratio of < 0.7 at screening.
2. Has clinical evidence of active infection, including, but not limited to, bronchitis, pneumonia, sinusitis, urinary tract infection, and cellulitis.
3. Has a history of malignancy within the last 2 years with the exception of basal cell carcinoma, chronic lymphocytic leukaemia (under observation) and prostate cancer requiring anti-androgens, localised treatment (minor surgery, radiotherapy) and/or managed by observation, and squamous cell carcinoma if diagnosed and successfully treated more than 6 months prior to the study. SCC diagnosed with the past 6 months will be exclusionary.
4. Patients experiencing cerebral hemorrhage or cerebral infarction at screening/baseline.
5. Has any condition other than IPF that, in the opinion of the investigator, is likely to result in the death of the subject within the next 2 years.
6. Presence of other disease that may interfere with testing procedures or in the judgement of the Investigator may interfere with trial participation or may put the patient at risk when participating in this trial.
7. Is likely to receive lung transplantation within the next 12 months.
8. Currently receiving high dose corticosteroid, cytotoxic (e.g., chlorambucil, azathioprine, cyclophosphamide, methotrexate), vasodilator therapy for pulmonary hypertension (e.g., bosentan), and or investigational therapy for idiopathic pulmonary fibrosis (IPF) or administration of such therapeutics within 4 weeks of initial screening (or 5 half-lives, whichever is longer). A current dose of less than or equal to 15 mg/day of prednisone or its equivalent is acceptable if the dose is anticipated to remain stable during the study.
9. Has a history of unstable or deteriorating cardiac or pulmonary disease (other than IPF) within the previous six months, including, but not limited to, the following:

   1. Unstable angina pectoris or myocardial infarction, or percutaneous coronary intervention within the last 6 months,
   2. Congestive heart failure requiring hospitalization,
   3. Uncontrolled clinically significant arrhythmias.
10. If female, the subject is pregnant or lactating or intending to become pregnant before participating in this study during the study and within (5 half- lives plus 30 days) after last dose of the study drug; or intending to donate ova during such time period.
11. Women considered to be of childbearing potential who do not use highly effective birth control methods during the study.
12. Known or suspected allergy to the trial drug or the relevant drugs given in the trial.
13. Involvement in a clinical research study within 4 weeks prior to screening and/or prior enrollment in the study. Participation in registry studies is permitted.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
A ≥50% reduction in the average number of coughs per hour over 24 hours comparing baseline to treatment period using an ambulatory cough monitor | Baseline and week 12 (≥11 weeks of treatment)
No worsening of force vital capacity (FVC) in either mL or % predicted | Baseline and week 12 (≥11 weeks of treatment)

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (4):
  - Vale Medical Practice, Brookvale, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Cairns Hospital, Cairns, Queensland
- New Zealand (2):
  - The University of Otago, Christchurch, Canterbury
  - Waikato Hospital, Hamilton, Waikato Region

IPD SHARING:
Plan to Share IPD: No